CLINICAL TRIAL: NCT06458933
Title: A Randomized Controlled Trial Testing Sage: A Couple Intervention for Borderline Personality Disorder
Brief Title: Testing Interventions for Borderline Personality Disorder.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: York University (Other)
Collaborators: Centre for Addiction and Mental Health (Other); Toronto Metropolitan University (Other); University of Windsor (Other); Kennesaw State University (Other); University of Winnipeg (Unknown); The Sashbear Foundation (Unknown)
Responsible Party: Principal Investigator, Skye Fitzpatrick, Associate Professor, York University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 495689
Record Dates: First submitted 2024-05-23; First posted 2024-06-14 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline Personality Disorder; Relationship dysfunction; Couple therapy; Emotion dysregulation
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sage (Experimental): Immediately receives 12 sessions of a couple psychotherapy designed to treat borderline personality disorder (BPD) and enhances relationship functioning simultaneously.
  Interventions: Behavioral: Sage
- SIP (Active Comparator): Immediately receives 12 individual sessions each (12 for people with borderline personality disorder (BPD), 12 for partners) of Supportive Individual Psychotherapy (SIP).
  Interventions: Behavioral: Supportive Individual Psychotherapy

INTERVENTIONS:
Behavioral: Sage — Sage is a 12-session manualized weekly intervention delivered to people with borderline personality disorder (BPD) and their intimate partners. The Sage intervention consists of three phases: Phase 1, orientation and safety which focuses on targeting destructive behaviours (e.g., suicide attempts and self harm engagement) by providing couples with safety strategies that target suicide risk/ crisis, education about BPD, the role of emotion dysregulation and intimate relationship dysfunction in maintaining it (~three sessions). Next, Phase 2, communication and emotion skills entails couples learning communication skills and strategies for identifying, expressing, and regulating emotions (~five sessions). Lastly, in Phase 3, cognitive skills and intervention termination, couples learn strategies to target negative cognitions that elicit emotion dysregulation and intimate relationship dysfunction (~four sessions).
  Arms: Sage
Behavioral: Supportive Individual Psychotherapy — Supportive Individual Psychotherapy (SIP) is a comparator in our control condition reflects enhanced usual care (i.e., supportive psychotherapy) for people with BPD. Both people with BPD and partners will receive SIP sessions separately over the course of 12 sessions, delivered by therapists. For both members of the couple, SIP will involve 12 sessions of a specific form of supportive psychotherapy based on client-centered, humanistic principles. This intervention involves creating a supportive therapeutic relationship, expressing empathy, and helping individuals feel understood. The SIP intervention is designed to support individuals in exploring their relationships and communication patterns as well as following the client's lead on what they want to work on.
  Arms: SIP

SUMMARY:
Borderline personality disorder (BPD) is a life-threatening, costly public health crisis affecting ~1-3% of North Americans, with 10% dying by suicide and annual healthcare costs of ~$63k (Canadian Dollars)/patient. Further, people with BPD's intimate relationships are highly disrupted, and their partners report elevated mental health problems but little access to treatment. Existing BPD treatments are resource-heavy, inaccessible, and 47% of people with BPD do not respond to them. These treatments also neglect relationship problems and intimate partner's mental health concerns, even though they are thought to play a key role in BPD maintenance. BPD interventions may produce stronger, quicker, and more durable outcomes if they incorporated partners to target both the emotional and relationship core of BPD. Moreover, incorporating partners into interventions may improve relationship outcomes and partner mental health without added resource investments.

Accordingly, members of our team developed Sage. Named after a plant that thrives in relationship with its ecosystem, Sage is a brief, 12-session conjoint intervention for people with BPD and their intimate partners that targets BPD, relationship conflict, and partner mental health. Our recent uncontrolled trial provides preliminary support for its efficacy.

As a next step in testing Sage, it is critical to utilize a Randomized Controlled Trial (RCT) design to identify if Sage is more efficacious than standard care that these couples typically receive; supportive individual psychotherapy (SIP) for people with BPD and their partners. The investigators propose to conduct the first RCT of Sage for couples wherein one member has BPD. The study will examine if Sage is more efficacious than SIP in improving BPD symptoms (primary outcome), as well as relationship conflict and partner mental health (secondary outcomes), as well as a range of other outcomes, from pre- to post-intervention, and post-intervention to follow-up. It will also investigate factors that influence treatment response, BPD severity, and related problems.

Up to 152 couples wherein one member has BPD will be randomized to receive Sage or SIP. Gold-standard measures of primary, secondary, and exploratory outcomes will be administered at baseline, mid-intervention, post-intervention, and a one-month, three- month, and six-month follow-up.

ELIGIBILITY:
INCLUSION CRITERIA

1. Participant with borderline personality disorder (BPD) meets full diagnostic criteria for BPD (i.e., five or more BPD diagnostic criteria per the Diagnostic and Statistical Manual of Mental Disorders-5-TR)
2. Both members are at least 19-years-old
3. Both members consent to study participation
4. Both members consent to a member of the research team contacting one of their provided emergency contacts if there are imminent safety concerns.
5. Both members consent to having assessment interviews and treatment sessions audio- and video-recorded
6. Both members members reside in Ontario (with no plan to leave the province during the course of the study)
7. Both members members are fluent in English
8. Both members are willing to receive emails about the study
9. Both members have regular internet access from a private location for completion of study appointments

EXCLUSION:

1. Severe intimate partner violence in their relationship in the past year (Endorsement of severe intimate partner violence items on Conflict Tactics Scale-2)
2. DSM-5 criteria A and B of schizophrenia, not better accounted for by BPD
3. Hospitalization in the past year for mania, or mania in the past three months
4. A substance/alcohol use disorder that is likely to require medical intervention (e.g., detoxification) to reduce use
5. A medical condition that is likely to require hospitalization within the next year
6. Scaled score below 70 on the Test of Premorbid Functioning, suggesting impaired intelligence and/or probable traumatic brain injury
7. Either participant in the dyad is not able to show proof of identification upon request at any point throughout the study or is not able to provide an accurate phone number or address upon request.
8. The individual with BPD is currently receiving an empirically-supported BPD treatment and is unwilling to pause the therapy for the duration of the active treatment phase

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-03-30 (Estimated)

PRIMARY OUTCOMES:
Zanarini Rating Scale for BPD (ZAN-BPD) | It will be administered only to people with BPD at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Interview measure of BPD severity. Scores range from 0 to 36, with higher scores reflecting higher severity of BPD symptoms.

SECONDARY OUTCOMES:
Conflict Resolution Scale | It will be administered people with BPD and partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of relationship conflict. Scores range from 0 to 52, with higher scores reflecting higher levels of conflict resolution.
Depression, Anxiety, and Stress Scale- depression subscale (partners) | It will be administered only to partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of depression. Scores range from 0 to 21, with higher scores reflecting higher levels of depression.
Generalized Anxiety Disorder 7 (GAD-7) | It will be administered only to partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of anxiety. Scores range from 0 to 21, with higher scores reflecting higher levels of anxiety.
Difficulties in Emotion Regulation Scale (DERS) | It will be administered only to partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of emotion dysregulation. Scores range from 36 to 180, with higher scores reflecting higher levels of emotion dysregulation.
Addiction Severity Index | It will be administered only to partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of problematic alcohol or substance use. Scores vary across substances and items, but higher scores indicate higher levels of problematic substance use.
Kessler Psychological Distress Scale-10 | It will be administered only to partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of psychological distress. Scores range from 10 to 50, with higher scores reflecting higher levels of psychological distress.

OTHER OUTCOMES:
Suicide Attempt Self-Injury Interview-modified | It will be administered only to people with BPD at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Interview measure of frequency of self-injury and suicidal behaviours. Scores reflect the frequency of suicidal and self-injurious behaviour.
Borderline Symptom List- 23 | It will be administered only to people with BPD at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of BPD severity. Scores range from 0 to 92, with higher scores reflecting higher levels of BPD severity.
Positive and Negative Affect Schedule (PANAS)- select subscales | It will be administered people with BPD and partners at baseline (pre-intervention), half-way through intervention, immediately after the intervention, and one, three, and six months after the intervention.
  Self-report measure of anger, fear, guilt, sadness, fatigue, positive emotion, negative emotion. Score ranges vary across subscales, with higher scores reflecting higher levels of emotion.
Communication Patterns Questionnaire-23 item version | It will be administered people with BPD and partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of communication patterns
Borderline Symptom List- 23-INFORMANT REPORT | It will be administered only to partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Informant-report measure of BPD severity Scores range from 0 to 92, with higher scores reflecting higher levels of partner's BPD severity.
Humor Styles Questionnaire - affiliative subscale | It will be administered people with BPD and partners at baseline (pre-intervention), 12 weeks, and 36 weeks.
  Self-report measure of humour and positive communication qualities. Scores range from 8 to 56, with higher scores reflecting higher levels of humour.
Perceived Relationship Quality Component | It will be administered people with BPD and partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of relationship satisfaction. Score ranges vary across subscales, with higher scores reflecting higher relationship quality.
Couples Satisfaction Inventory- 16 item version | It will be administered people with BPD and partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of relationship satisfaction. Scores range from 0 to 81, with higher scores reflecting higher levels of relationship satisfaction.
Sage skills use measure | It will be administered people with BPD and partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Use of Sage skills self-report measure, created for present study. Scores range from 0 to 60, with higher scores reflecting higher levels of Sage skill use.
Sage skills use measure (in session) | It will be administered to people with BPD and partners in the Sage condition at the beginning of every session.
  Use of Sage skills self-report measure, created for present study. Scores reflect the number of times a skill was used.
Feinberg Brief Co-Parenting Scale | It will be administered people with BPD and partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of co-parenting experiences. Scores range from 0 to 72, with higher scores reflecting higher levels positive co-parenting.
Empathic accuracy measure | It will be administered people with BPD and partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self and informant-report measure of one's own and one's partner's emotions. Scores for each emotion range from 1 to 5, with higher scores indicating higher levels of emotion.
Working Alliance Inventory- Short form | It will be administered to people with BPD and partners, as well as their therapists, approximately weekly from weeks one to 12.
  Self-report measure of working therapeutic alliance. Scores range from 12 to 60, with higher scores reflecting a stronger therapeutic alliance.
Posttraumatic Checklist-5 (PCL-5) | It will be administered people with BPD and partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of PTSD symptoms. Scores range from 0 to 80, with higher scores reflecting higher levels of PTSD severity.
Informant Difficulties in Emotion Regulation Scale (DERS) | It will be administered people with BPD and partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Informant-report measure of emotion dysregulation. Scores range from 8 to 40, with higher scores reflecting higher levels of informant-reported emotion dysregulation.
Depression, Anxiety, and Stress Scale- depression subscale (people with BPD) | It will be administered only to people with BPD at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of depression. Scores range from 0 to 21, with higher scores reflecting higher levels of depression.
Generalized Anxiety Disorder 7 (GAD-7) | It will be administered only to people with BPD at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of anxiety. Scores range from 0 to 21, with higher scores reflecting higher levels of anxiety.
Difficulties in Emotion Regulation Scale (DERS) | It will be administered only to people with BPD at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of emotion dysregulation. Scores range from 36 to 180, with higher scores reflecting higher levels of emotion dysregulation.
Experiences of Shame Scale | It will be administered only to people with BPD at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of shame. Scores range from 25 to 100, with higher scores reflecting higher levels of shame.
Impulsive Behaviour Scale | It will be administered only to people with BPD at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of impulsive behaviour. Scores range from 25 to 125, with higher scores reflecting higher frequency of impulsive behaviour.
Self Compassion Scale-Short form | It will be administered people with BPD at baseline (pre-intervention), 12 weeks, and 36 weeks.
  Self-report measure of self-compassion Scores range from 12 to 60, with higher scores reflecting higher levels of self-compassion.
Multidimensional scale of perceived social support | It will be administered people with BPD and partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of perceived social support. Scores range from 1 to 7, with higher scores reflecting higher levels of perceived social support.
Sexual functioning and satisfaction items | It will be administered people with BPD and partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Singular items measuring sexual functioning and satisfaction. Higher scores generally reflect higher sexual satisfaction or frequency of sexual activity.
Break up items | It will be administered people with BPD and partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Singular items measuring whether the relationship has ended.
Conflict tactics scale-2: Negotiation subscale | It will be administered people with BPD and partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of negotiation communication. Scores range from 0 to 36, with higher scores reflecting higher levels negotiation communication.
Subjective emptiness scale | It will be administered only to people with BPD at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of emptiness. Higher scores reflect higher emptiness.
Inventory of Interpersonal Problems (IIP)- BPD subscale | It will be administered only to people with BPD at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of interpersonal problems in BPD. Scores range from 0 to 72, with higher scores reflecting higher levels of interpersonal problems.
Addiction Severity Index | It will be administered only to people with BPD at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of problematic alcohol or substance use. Scores vary across substances and items, but higher scores indicate higher levels of problematic substance use.
Kessler Psychological Distress Scale-10 | It will be administered only to people with BPD at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of psychological distress. Scores range from 10 to 50, with higher scores reflecting higher levels of psychological distress.
Brief Inventory of Psychosocial Functioning | It will be administered people with BPD and partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of social functioning. Scores range from 0 to 44, with higher scores reflecting more difficulties in social functioning.
Short Form (12) Health Survey | It will be administered people with BPD and partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of health
Barratt Impulsiveness Scale-11 | It will be administered only to people with BPD at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of impulsivity
Columbia Suicide Severity Rating Scale- Suicidal Ideation section | It will be administered only to people with BPD at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Interview measure of suicidal ideation. The presence and intensity of suicidal ideation are scored separately and range from 0 to 5 and 0 to 25, respectively, with higher scores reflecting higher severity.
Dissociative Experiences Scale II | It will be administered only to people with BPD at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of dissociation. Higher scores reflect higher levels of dissociation.
Mental Health Utilization | It will be administered only to people with BPD at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Qualitative interview of measure of mental health service utilization.
Emergency Department Visits | It will be administered only to people with BPD at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Interview of measure of frequency of emergency department visits and reasons for them.
World Health Organization Quality of Life Items | It will be administered people with BPD and partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Three items measuring health, physical functioning, quality of life. Scores range from 1 to 5, with higher scores reflecting higher perceived health, work functioning or quality of life.
Revised University of California-Los Angeles Loneliness Scale | It will be administered people with BPD and partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of loneliness Scores range from 20 to 80, with higher scores reflecting higher levels of loneliness.
Emotion Regulation Questionnaire | It will be administered people with BPD and partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Measure of suppression and reappraisal emotion regulation strategy use. Scores range from 4 to 28 for suppression, and 6 to 42 for reappraisal, with higher scores reflecting higher emotion regulation strategy use.
Relationship Questionnaire | It will be administered people with BPD and partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  4-item measure of attachment. Each attachment style is rated on a scale from 1 to 7, with higher scores reflecting a higher measure of each attachment style.
Mentalization Scale | It will be administered people with BPD and partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of mentalization. Scores range from 28 to 140.
Interpersonal Needs Questionnaire | It will be administered people with BPD and partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of perceived burdensomeness and thwarted belongingness. Higher scores reflect higher levels of perceived burdensomeness and thwarted belongingness.
Test of Roles and Reactions in Dyads (TORRID) | It will be administered only to partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of roles partners of people with BPD play and their experiences in their relationship. Scores range depending on subscale, with higher scores reflecting higher identification with the role in question.
Burden assessment scale | It will be administered only to partners at baseline (pre-intervention), six weeks, 12 weeks, 16 weeks, 24 weeks, and 36 weeks.
  Self-report measure of burden. Score ranges vary across subscales, with higher scores reflecting higher levels of burden.
The Satisfaction With Therapy and Therapist Scale-Revised (STTS-R) | It will be administered to people with BPD and partners at immediately after the intervention (12 weeks).
  Self-report measure of satisfaction with intervention and therapist. Scores range from 12 to 60, with higher scores reflecting higher levels of satisfaction with intervention and therapist.
Behavioural communication sample | It will be administered to people with BPD and their partners in the Sage condition only at the first and last intervention session.
  A videorecording of the couple discussing a problem in their relationship. The sample is then coded using a reliable and valid coding system for adaptive and maladaptive communication behaviours.

CONTACTS AND LOCATIONS:
Locations (1):
- York University, Toronto, California, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be posted on a public, online data repository for the purpose of sharing it with the broader scientific community, to promote integrity and transparency in our research and allow other researchers to replicate our results from an open science framework.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Following publication of primary study outcomes